CLINICAL TRIAL: NCT03494660
Title: A Longitudinal Outcomes Study of the Subchondroplasty® Procedure in the Hip
Brief Title: SCP Hip Outcomes Study
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CSU2017-03KC
Record Dates: First submitted 2018-04-03; First posted 2018-04-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Subchondral Cysts; Subchondral Bone Edema; Bone Marrow Edema; Insufficiency Fractures; Avascular Necrosis of Hip; Femoroacetabular Impingement; Dysplasia; Hip
Keywords: Subchondroplasty; Bone Marrow Lesion; Arthroscopy; Bone Substitute Material; AccuFill; Subchondral Bone Defect
MeSH Terms: conditions — Bone Cysts; Fractures, Stress; Femoracetabular Impingement; Hip Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Subchondroplasty Procedure with AccuFill — Injection of the commercially available flowable calcium phosphate (CaP) synthetic bone-void filler, AccuFill®, into subchondral bone defects in the hip (Subchondroplasty (SCP) Procedure).

SUMMARY:
Post-market clinical outcomes study to collect data on the short- and long-term outcomes for subjects who are undergoing or have undergone the Subchondroplasty® (SCP®) Procedure in the hip in a standard clinical setting. Outcomes to be assessed include medication usage, pain, function, activity levels and patient satisfaction.

DETAILED DESCRIPTION:
This study is designed as a post-market, single arm, non-randomized multi-center investigation.

Male and female subjects, at least 18 years of age, with at least one subchondral bone defect in the form of a cyst and/or bone marrow lesion (BML), insufficiency fracture or bone defect associated with early stage avascular osteonecrosis (AVN) in the femoral head, femoral neck and/or acetabulum who are suitable candidates for use of AccuFill during the Subchondroplasty Procedure are eligible for enrollment in this study.

A maximum of 15 study sites, in the United States of America, will enroll a target of 50 subjects.

Each Investigator must obtain IRB approval, or favorable opinion by an EC, prior to consent of the first subject; no study-related procedures can occur without the approval and oversight of a registered IRB or EC. If the study site does not have an IRB of record, a central IRB may be utilized upon approval by Zimmer Biomet.

Demographics, medical history, hip history and use of pain medication and therapy will be recorded at the time of subject consent. Additionally, patient reported outcomes measures will be obtained pre-operatively. Operative details including the SCP Procedure, concomitant surgical procedures and intraoperative safety events will be recorded at the time of surgery. Prospective subjects will be considered enrolled in this study once their Subchondroplasty Procedure has been performed.

Subjects will complete only the Numeric Pain Scale at 2 weeks post-operatively. Thereafter, subjects will complete self-reported outcomes measures post-operatively at 6 weeks, 12 weeks, 6 months, 1 year and 2 years. These measures include information on pain medication and therapy, pain levels, function, activity and subject satisfaction. Screening for adverse events and conversion will occur throughout the study.

Subjects will complete the study at 2 years or will be withdrawn if they undergo conversion of the Subchondroplasty site. For the purposes of this protocol, a conversion will be defined as total hip arthroplasty or any procedure involving removal of the AccuFill material on the index hip.

ELIGIBILITY:
Inclusion Criteria:

* Candidates must meet ALL of the following:

  1. Surgeon considers the patient appropriate for the SCP Procedure of the hip.
  2. Subchondral bone defect(s) in the femoral head, femoral neck and/or acetabulum has been confirmed via radiographic finding on MRI or x-ray.
  3. Subject provides voluntary signature on the IRB approved Informed Consent Form.
  4. Subject is at least 18 years of age.
  5. Subject must be physically and mentally willing and able, in the Investigator's opinion at the time of enrollment, to be compliant with the protocol and complete outcome forms via email, telephone, in-person or by regular mail.

Exclusion Criteria:

* Candidates will be excluded if they meet ANY of the following:

  1. Subject has collapse of subchondral bone.
  2. Subject is pregnant at the time of surgery.
  3. Subject is incarcerated.
  4. Subject is involved in active litigation related to the condition being treated.
  5. Subject is not comfortable with speaking, reading, and understanding questions and providing responses in an available language for the PROs in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 50 subjects, each with at least one subchondral bone defect in the form of a cyst and/or bone marrow lesion (BML), insufficiency fracture or bone defect associated with early stage avascular osteonecrosis (AVN) in the femoral head, femoral neck and/or acetabulum who are suitable candidates for use of AccuFill during the Subchondroplasty Procedure are eligible for enrollment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2024-10-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Harris Hip Score (mHHS) from baseline at 12 months | 12 months
  Change in Modified Harris Hip Score using a 0-100 overall score, from baseline at 12 months. Subscales of pain, function, and activity levels are combined to generate the overall score. Pain is scored out of 44 possible points, function is scored out of 33 possible points and subject activities are scored out of 14 possible points. The maximum score of 91 is multiplied by 1.1 to give a total score out of 100; a higher score represents better patient reported pain, function and activity levels.

SECONDARY OUTCOMES:
Incidence and severity of device and/or procedure related adverse events and surgical conversions | 2 years
  Summary and description of procedure and device related adverse events and surgical conversions and relatedness to the bone substitute material and procedure
Change in numeric pain score from baseline at 12 months | 12 months
  Change in numeric pain score using a 0-10 scale, from baseline at 12 months. Patient's current hip pain will be selected where 0 describes no pain and 10 describes worst possible pain on average over the past 24 hours.
Change in Hip Outcome Score from baseline at 12 months | 12 months
  Change in patient Activities of Daily Living and Sports, from baseline at 12 months.
  The Activities of Daily Living (ADL) and Sports subscales are scored separately. On the ADL subscale, the score on each of the items are added together to get the item score total. The total number of items with a response is multiplied by 4 to get the highest potential score. If the subject answers all 17 items, the highest potential score is 68. If one item is not answered the highest score is 64, if two are not answered the total highest score is 60, etc. The item score total is divided by the highest potential score. This value is then multiplied by 100 to get a percentage.
  The Sports subscale is scored in a similar manner with the highest potential score being 36. A higher score represents a higher level of physical function for both the ADL and Sports subscales.
Change in EuroQol-5 Dimensions (EQ-5D) from baseline at 12 months | 12 months
  Change in patient quality of life from baseline at 12 months. A scoring function is created using a population preference weighted health index.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Eisenhower Desert Orthopedic Center, Rancho Mirage, California
  - Andrews Research & Education Foundation, Gulf Breeze, Florida
  - OrthoIllinois, Rockford, Illinois
  - University of Kentucky Research Foundation, Lexington, Kentucky
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Subchondroplasty® (SCP®) Procedure — http://subchondroplasty.com/